CLINICAL TRIAL: NCT05492903
Title: Translating an Intervention to Address Chronic Pain Among Home Care Workers
Brief Title: COMmunity of Practice And Safety Support for Navigating Pain (COMPASS-NP)
Acronym: COMPASS-NP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Ryan Olson, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: e20412
Record Dates: First submitted 2022-02-18; First posted 2022-08-09 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Pain Management; Ergonomics; Wounds and Injuries
Keywords: injury prevention; pain management; ergonomics; home care workers; total worker health; cognitive behavioral therapy
MeSH Terms: conditions — Agnosia; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: cluster-randomized waitlist control design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention during weeks 0-10 (10 weekly group sessions). Follow-up with no treatment during weeks 11-20.
  Interventions: Behavioral: COMmunity of Practice And Safety Support for Navigating Pain (COMPASS-NP)
- Waitlist Control (Other): Usual practice during weeks 0-10. Intervention during weeks 11-20 (10 weekly group sessions).
  Interventions: Behavioral: COMmunity of Practice And Safety Support for Navigating Pain (COMPASS-NP)

INTERVENTIONS:
Behavioral: COMmunity of Practice And Safety Support for Navigating Pain (COMPASS-NP) — A peer-led and supportive group program (10 weekly sessions) designed to address the needs of HCWs with chronic or elevated pain. The intervention will integrate work-based injury protections with pain education and cognitive-behavioral therapy strategies for pain self-management.

SUMMARY:
Home care workers (HCWs) are at-risk for chronic pain and associated problems, including emotional distress, opioid use and misuse, and work-related disability. To address these issues, the proposed study will adapt an established peer-led and supportive group program to address the needs of HCWs with chronic pain. The new program, named COMPASS for Navigating Pain (COMPASS-NP), will integrate work-based injury protections with pain education and cognitive-behavioral therapy strategies for pain self-management in order to reduce pain interference with HCWs' work and life, and advance their safety, health, and well-being.

DETAILED DESCRIPTION:
Organizational intervention research can be all breakthrough with no follow-through. Few effective interventions developed by scientists are widely adopted in practice. To address this research-to-practice gap and address a socially important problem, the investigators will translate their established and disseminated COMPASS (COMmunity of Practice And Safety Support) intervention to address the needs of home care workers (HCWs) with chronic pain. The burden of injuries and pain is great among HCWs, which places them at-risk for emotional distress, opioid use/misuse, and work-related disability. Moreover, HCWs are predominantly low income, middle aged women. Between 1999 and 2015 middle-aged women experienced a 471% increase in prescription opioid-related overdoses. COMPASS is a peer-led and scripted group curriculum that produced many significant impacts on meaningful outcomes for HCWs in a randomized controlled trial (Cohen's d range = .45 to .84), including increased safety communication with clients and hazard correction in homes. COMPASS was subsequently adopted by the Oregon Home Care Commission, and is currently offered statewide as a paid training course to publicly funded HCWs. While these are exceptional research-to-practice impacts, the original curriculum did not directly address chronic pain, and resulted in only small non-significant reductions in pain severity. The investigators also found that HCWs with pain-related limitations at baseline made significant safety changes, but experienced less benefit from the intervention than workers without limitations. An added barrier is that protective low-tech ergonomic tools (e.g., slide boards, transfer belts) are typically not funded by insurance. The investigators' qualitative research revealed that low-wage HCWs are often forced to improvise or do without such tools. In the translation plan, existing COMPASS lessons will be adapted for HCWs with chronic pain, and new lessons from the Pain Survival Guide (co-authored by Dr. Turk, Co-I) will integrate pain education and proven cognitive-behavioral therapy pain self-management strategies. The investigators will also strengthen injury protections by including an online ergonomic assessment and voucher for HCWs to purchase tools. The translated COMPASS for Navigating Pain (COMPASS-NP) intervention will be evaluated with a cluster randomized waitlist control design. The primary hypothesis is that COMPASS-NP will reduce pain interference with work and life. Secondary outcomes include pain/injury prevention behaviors (e.g., ergonomic tool use), injuries, pain severity, risk for opioid misuse, and worker well-being. Regional implementation and evaluation with partners in Oregon (government), Washington (labor), and Idaho (private sector) will maximize dissemination knowledge and impact. The 5-year project will accomplish 4 aims: 1) Adapt and pilot COMPASS-NP in Oregon; 2) Determine effects of COMPASS-NP across Oregon, Washington, and Idaho; 3) Describe the translation and implementation of COMPASS-NP across partners and systems; and 4) Disseminate COMPASS-NP knowledge, tools, and toolkits.

ELIGIBILITY:
Inclusion Criteria:

* 18 years (adults)
* Employed as a home care worker
* Has chronic pain (pain lasting 3+ months and > 4 average intensity)
* The presence of pain interference with work (response of 'agree' or 'strongly agree' on single-item)
* Currently working 4 hours or more per week
* Access to the internet with a video capable device (e.g., smart phone, tablet, or computer)

Exclusion Criteria:

* Prior exposure to the original COMPASS program
* Experiencing a surgery in the prior 6 months
* Current pregnancy or intention to become pregnant during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Between Groups Difference in Changes in Ratings of Pain Interference with Work | Changes between 0 weeks and 10 weeks
  Work Limitations Questionnaire (1-5; 5=worst [limited all the time]). Assesses limitations related to time, physical, mental-interpersonal, and outputs.
Between Groups Difference in Changes in Ratings of Pain Interference with Life | Changes between 0 weeks and 10 weeks
  Brief Pain Inventory Subscale on pain interference (0-10; 10=worst [completely interferes]). Interference related to general activity, walking, work, relations with other people, sleep, and enjoyment of life.

SECONDARY OUTCOMES:
Between Groups Difference in Changes in Reported Number of Pain/Injury Prevention Actions | Changes between 0 weeks and 10 weeks
  Assessment questions developed by authors addressing total number of safety actions taken during the prior 10 weeks (0 to 5 or more; 0=worst [no actions taken]). Sum of counts for five items that address new ergonomic tool use or techniques for moving objects or assisting client mobility; new ergonomic tools or techniques for housekeeping; correcting slip, trip, and fall hazards in homes; correcting "other" hazards in homes; and talking with client about improving safety.
Between Groups Difference in Changes in Reported Number of Minor Injuries | Changes between 0 weeks and 10 weeks
  Question developed by authors addressing the number of minor injuries (minor cuts, bruises, back/neck pain or sprains) during the previous 10 weeks (5 or more=worst [highest possible number of reported minor injuries).
Between Groups Difference in Changes in Reported Number of Lost Work Time Injuries | Changes between 0 weeks and 10 weeks
  Question developed by authors addressing the number of injuries resulting in one or more days off of work during the prior 10 weeks (0-5 or more lost work time injuries; 5 or more=worst [highest possible reported number of injuries).
Between Groups Difference in Changes in the Rating of Average Pain Severity | Changes between 0 weeks and 10 weeks
  Brief Pain Inventory item addressing average pain severity, with author-selected time anchor of during the past week (0-10; 10=worst [worst pain possible]).
Between Groups Difference in Changes in Ratings of Well-being | Changes between 0 weeks and 10 weeks
  Patient-Reported Outcomes Measurement Information System (PROMIS) Global-Mental Health Subscale (items 2,4, and 5 are rated 5-1; 1=worst [poor]; item 10 is rated 1-5 and reverse coded; before reverse coding 5=worst [always bothered]). Items assess quality of life, mental health and mood/thinking, satisfaction with social relationships, and emotional problems.
Between Groups Difference in Changes in Daily Minutes of Physical Activity | Changes between 0 weeks and 10 weeks
  Actigraphy sample of seven days (hip-worn) will be collected to calculate average daily minutes of physical activity (focused on combined light and moderate intensity minutes).
Between Groups Difference in Changes in Average Nightly Sleep Duration | Changes between 0 weeks and 10 weeks
  Actigraphy sample of seven days (wrist-worn) will be collected to calculate average hours and minutes of sleep duration for the main sleep period each night.
Between Groups Difference in Changes in Average Nightly Sleep Efficiency | Changes between 0 weeks and 10 weeks
  Actigraphy sample of seven days (wrist-worn) will be collected to calculate average sleep efficiency (percent of time in bed spent asleep) for the main sleep period.
Between Groups Difference in Changes in Pain Medication Use | Changes between 0 weeks and 10 weeks
  Brief Pain Inventory item assessing frequency of pain medication use per 24 hours. Five frequency interval options range from "not every day" to "more than 6 times per day" (more than 6 is worst [highest daily frequency]).
Between Groups Difference in Changes in Risk of Future Opioid Misuse | Changes between 0 weeks and 10 weeks
  Screener and Opioid Assessment for Patients with Pain-Revised (SOAPP-R; for workers not currently using opioids). Item ratings of 0-4 (4=worst [very often]) with a total sum of 18 indicating positive for being at-risk for future opioid misuse.
Between Groups Difference in Changes in Current Opioid Misuse | Changes between 0 weeks and 10 weeks
  Current Opioid Misuse Measure (COMM; for workers currently using opioid medications). Ratings of 0-4 (4=worst [very often]) with a score of 9 or greater indicating a positive for current opioid misuse.

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Olson R, Hess JA, Turk D, Marino M, Greenspan L, Alley L, Donovan C, Rice SPM. COMMunity of Practice And Safety Support for Navigating Pain (COMPASS-NP): study protocol for a randomized controlled trial with home care workers. Trials. 2023 Apr 10;24(1):264. doi: 10.1186/s13063-023-07149-8. PMID 37038235